CLINICAL TRIAL: NCT02231307
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Clinical Efficacy and Safety of SUBLIVAC FIX Birch Immunotherapy in Patients Suffering From Allergic Rhinitis/Rhinoconjunctivitis Caused by Birch Pollen.
Brief Title: SUBLIVAC FIX Birch Phase III Short-term Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB/0042
Record Dates: First submitted 2014-08-25; First posted 2014-09-04 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Birch Pollen Induced Rhinitis/Rhinoconjunctivitis
Keywords: sublingual immunotherapy; birch pollen; allergic rhinitis / rhinoconjunctivitis; efficacy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUBLIVAC FIX Birch 0 AUN/ml (Placebo Comparator)
  Interventions: Drug: SUBLIVAC FIX Birch
- SUBLIVAC FIX Birch 40,000 AUN/ml (Experimental)
  Interventions: Drug: SUBLIVAC FIX Birch

INTERVENTIONS:
Drug: SUBLIVAC FIX Birch

SUMMARY:
The aim of this phase III study is to asses if SUBLIVAC FIX Birch is safe and effective in reducing birch allergy induced symptoms and birch allergy medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 and ≤65 years
* Moderate-to-severe birch pollen induced allergic rhinitis/rhinoconjunctivitis based on ARIA classification for at least 2 consecutive years
* FEV1 (forced expiratory volume at one second) > 70% (of predicted value) for patients with a history of asthma, FEV1 > 70% or PEF (peak expiratory flow) > 80% (of predicted value) for patients without a history of asthma
* Positive SPT (skin prick test) for birch pollen (mean wheal diameter ≥ 3mm compared to negative control; negative control should be negative; histamine control should be positive (mean wheal diameter ≥ 3mm)) assessed during screening.
* Serum specific anti-birch IgE (immunoglobulin E) concentration >0.7 U/ml
* Patients should be willing and capable to complete an e-diary daily during the birch pollen season (≥ 60% compliance in completion between Visit 1 and 2).
* A positive Nasal Provocation Test to birch pollen at Visit 2 (Lebel score ≥ 6) or a documented positive test within 1 year before start of treatment

Exclusion Criteria:

* Patients sensitized and symptomatic to pets should not be included if they are regularly exposed to pets
* Specific immunotherapy (SCIT or SLIT) with birch pollen or a cross-reacting allergen within the last 5 years
* SPT positive (mean wheal diameter ≥ 3mm compared to negative control; negative control should be negative; histamine control should be positive (mean wheal diameter ≥ 3mm)) patients to allergen(s) other than birch pollen, in the absence of a negative provocation test for this allergen(s) (within 1 year), who are expected to have clinically relevant symptoms during the birch pollen season
* Completed unsuccessful allergen-specific immunotherapy (SCIT or SLIT) within the last 5 years
* (Ongoing) allergen-specific immunotherapy (SCIT or SLIT) with any allergen(s) during the study period
* Vaccination one week before start of treatment and/or during the up-dosing phase
* Treatment with experimental products within the last 3 months or biologicals (including anti-IgE or TNF (tumor necrosis factor) - α treatment) within the last 6 months or during the study
* Uncontrolled asthma or other active respiratory diseases
* Clinically significant chronic sinusitis, ocular infection or severe inflammation of the oral mucosa
* Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
* Active malignancies or any malignant disease in the last 5 years
* Acute or chronic disease that in the opinion of the investigator is an additional risk for the patients, including but not limited to the following: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine disorders, clinically significant renal or hepatic diseases, or haematological disorders
* Diseases with a contra-indication for the use of adrenaline (e.g. hyperthyroidism, glaucoma)
* Use of systemic corticosteroids 4 weeks before the study
* Treatment with systemic or local β-blockers
* Known hypersensitivity to any of the excipients (Disodium phosphate dihydrate, Sodium dihydrogen phosphate dehydrate, aminocaproic acid, Peppermint oil, Caramel Colorant or Glycerol)
* A positive urine pregnancy test, lactation or inadequate contraceptive methods (adequate methods: oral contraceptives, IUD (intrauterine device), condom use and having no sexual relationship with a man)
* Alcohol-, drug or medication abuse
* Lack of co-operation or compliance
* Severe psychiatric, psychological, or neurological disorders
* Any physical or mental condition that precludes administration or allergen-specific immunotherapy, compliance or participation in a clinical trial
* Patients who are employees of the department, 1st grade relatives, or partners of the investigator
* Patients who have planned holidays outside the country for more than 7 continuous days during the defined pollen season (1st of March till 31st of May)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
combined symptom medication score | 3 months

SECONDARY OUTCOMES:
symptom score | 3 months
Quality of Life questionnaires | 3 months
Serum specific immunoglobulin levels | up to 9 months
local and systemic reactions | up to 9 months
(serious) adverse events | up to 9 months
blood safety parameters | up to 9 months
urinalysis | up to 9 months
medication score | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pfaar, Prof. Dr., Principal Investigator — Zentrum für Rhinologie und Allergologie, An-den-Quellen-10, 65189 Wiesbaden, Germany
Locations (40):
- Belgium (5):
  - Cliniques universitaire St. Luc, Brussels
  - University Hospital, Ghent
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
  - CHU de Liege, Liège
- Czechia (7):
  - AKI spol. s.r.o., Brno
  - Alergologicka ambulance, Břeclav
  - Alergologicka ambulance, Liberec
  - Ordinace Alergologie, Most
  - Respiral s.r.o., Pilsen
  - Ustav imunologie a alergologie, Pilsen
  - Kasmed s.r.o., Tábor
- Germany (10):
  - CIMS Studienzentrum Bamberg, Bamberg
  - Charite Universitatsmedizin, Berlin
  - Dermatologikum Hamburg, Hamburg
  - HNO Gemeinschaftspraxis, Heidelberg
  - Hautarztpraxis fur Dermatologie & asthetische medizin, Hildesheim
  - Praxis fur Atemwegserkrankungen, Leipzig
  - FA HNOW Allergologie, Saalfeld
  - Praxis Dr. Jager, Schwabach
  - Klinik fur Dermatologie & Allergologie, Stuttgart
  - HNO Wiesbaden Institute for Allergology and Rhinology, Wiesbaden
- Poland (13):
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bialystok
  - NZOZ ZLS Medex Sp. z o.o. Poradnia Alergologiczna, Bielsko-Biala
  - SP-ZOZ Osrodek Zdrowia w Bienkowce, Bieńkówka
  - NZOZ Clinica Vitae, Gdansk
  - Grazyna Pulka Specjalistyczny Osrodek 'All-Med', Krakow
  - NZOZ Centrum Alergologii Krzysztof Buczylko, Lodz
  - Poradnia Alergologii i Chorob Pluc Uniwersytecki Szpital Kliniczny, Lodz
  - NZOZ Centrum Alergologii, Lublin
  - Przychodnia Alergologiczno-Pulmonologiczna ALERGOPNEUMA, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - Centrumk Medyczne Lucyna i Andrzej Dymek, Strzelce Opolskie
  - ALERGOMED Specjalistyczna Przychodnia Lekarska, Tarnów
  - EMC Intytut Medyczny S.A. Przychodnia przy Lowieckiej, Wroclaw
- Slovakia (5):
  - ALIAN s.r.o. Ambulancia alergologie a klinickej imunologie, Bardejov
  - Alerso s.r.o. Imunoalergologicka ambulancie, Košice
  - STALERG s.r.o. Imunoalergologicka ambulancia, Košice
  - DANIMED, spol. s.r.o. Ambulancia klinkckej imunologie a alergologie, Levice
  - EMED s.r.o. Alergoimunologicke centrum, Prešov

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419
- [Derived] Pfaar O, Bachert C, Kuna P, Panzner P, Dzupinova M, Klimek L, van Nimwegen MJ, Boot JD, Yu D, Opstelten DJE, de Kam PJ. Sublingual allergen immunotherapy with a liquid birch pollen product in patients with seasonal allergic rhinoconjunctivitis with or without asthma. J Allergy Clin Immunol. 2019 Mar;143(3):970-977. doi: 10.1016/j.jaci.2018.11.018. Epub 2018 Nov 30. PMID 30508538